CLINICAL TRIAL: NCT02466269
Title: A Modified Preauricular Approach to Treat Diacapitular Condylar Fractures: The Supratemporalis Approach
Brief Title: Treatment of Diacapitular Condylar Fractures
Status: Completed | Type: Observational
Sponsor: Hui Li (Other)
Collaborators: West China College of Stomatology (Other)
Responsible Party: Sponsor-Investigator, Hui Li, Principal Investigator, West China College of Stomatology
Organization: West China College of Stomatology (Other)
Other Study IDs: hui_owen
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Mandibular Fractures
Keywords: Facial Nerve Injuries
MeSH Terms: conditions — Mandibular Fractures; Facial Nerve Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- the preauricular approach: A classic preauricular incision was used to treat diacapitular condylar fractures
  Interventions: Procedure: The supratemporalis approach

INTERVENTIONS:
Procedure: The supratemporalis approach — The supratemporalis approach was applied in treatment of diacapitular condylar fractures

SUMMARY:
A new surgical approach, denoted as the supratemporalis approach, was designed to treat diacapitular condylar fractures of the mandibular condyle.This approach prevented facial nerve injury and did not increase the frequency of other complications. Therefore, the investigators suggest this surgical procedure as a routine and safe approach to diacapitular condylar fractures, which can also be applied to temporomandibular joint（TMJ）and to the zygomatic arch.

DETAILED DESCRIPTION:
Eighty-four patients (112 sides) with diacapitular condylar fractures were treated surgically. Forty-four patients (64 sides) were treated with the supratemporalis approach, and forty patients (48 sides) were treated with traditional preauricular approach. Data on the surgical procedures and complications were recorded. The follow-up periods were 12 -24months. The evaluated parameters include facial nerve injury，the maximum mouth opening, mandibular movements, occlusion, scar formation，hemorrhage and infection.Seven patients sustained facial nerve paresis in the group treated with the traditional preauricular approach. No case of facial nerve injury was observed in the supratemporalis approach group. No other significant differences were detected between the two groups in the functional and esthetic aspects.

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiographical diagnosis of DFs;

Exclusion Criteria:

1. condylar fractures with undisplaced fractures;
2. Fractures without the reduction of the condylar height;
3. A obvious scar at the temporal region, affecting the placement of the original incision.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with diacapitular condylar fractures
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from facial nerve function at 24 hours postoperatively | 24 hours
  The patients were instructed to raise their eyebrows, wrinkle the forehead, gently close the eyes, blow the cheek and smile. Paralysis of the facial nerve was deemed to have occurred if these motions were not achieved.
Change from facial nerve function at 1 week postoperatively | 1 week
  The patients were instructed to raise their eyebrows, wrinkle the forehead, gently close the eyes, blow the cheek and smile. Paralysis of the facial nerve was deemed to have occurred if these motions were not achieved.
Change from facial nerve function at 3 months postoperatively | 3 months
  The patients were instructed to raise their eyebrows, wrinkle the forehead, gently close the eyes, blow the cheek and smile. Paralysis of the facial nerve was deemed to have occurred if these motions were not achieved.
Change from facial nerve function at 6 months postoperatively | 6 months
  The patients were instructed to raise their eyebrows, wrinkle the forehead, gently close the eyes, blow the cheek and smile. Paralysis of the facial nerve was deemed to have occurred if these motions were not achieved.
Change from facial nerve function at 12 months postoperatively | 12 months
  The patients were instructed to raise their eyebrows, wrinkle the forehead, gently close the eyes, blow the cheek and smile. Paralysis of the facial nerve was deemed to have occurred if these motions were not achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, DMD, Study Director — Department of Oral & Maxillofacial Surgery, West China Hospital of Stomatology, Sichuan University

REFERENCES:
- [Background] Amaratunga NA. A study of condylar fractures in Sri Lankan patients with special reference to the recent views on treatment, healing and sequelae. Br J Oral Maxillofac Surg. 1987 Oct;25(5):391-7. doi: 10.1016/0266-4356(87)90088-x. PMID 3478083
- [Background] Silvennoinen U, Iizuka T, Lindqvist C, Oikarinen K. Different patterns of condylar fractures: an analysis of 382 patients in a 3-year period. J Oral Maxillofac Surg. 1992 Oct;50(10):1032-7. doi: 10.1016/0278-2391(92)90484-h. PMID 1527654
- [Background] Chrcanovic BR, Abreu MH, Freire-Maia B, Souza LN. 1,454 mandibular fractures: a 3-year study in a hospital in Belo Horizonte, Brazil. J Craniomaxillofac Surg. 2012 Feb;40(2):116-23. doi: 10.1016/j.jcms.2011.03.012. Epub 2011 Mar 31. PMID 21458284
- [Background] Ellis E 3rd, Moos KF, el-Attar A. Ten years of mandibular fractures: an analysis of 2,137 cases. Oral Surg Oral Med Oral Pathol. 1985 Feb;59(2):120-9. doi: 10.1016/0030-4220(85)90002-7. No abstract available. PMID 3856795
- [Background] Marker P, Nielsen A, Bastian HL. Fractures of the mandibular condyle. Part 1: patterns of distribution of types and causes of fractures in 348 patients. Br J Oral Maxillofac Surg. 2000 Oct;38(5):417-21. doi: 10.1054/bjom.2000.0317. PMID 11010766
- [Background] Loukota RA, Eckelt U, De Bont L, Rasse M. Subclassification of fractures of the condylar process of the mandible. Br J Oral Maxillofac Surg. 2005 Feb;43(1):72-3. doi: 10.1016/j.bjoms.2004.08.018. PMID 15620780
- [Background] Lindahl L. Condylar fractures of the mandible. I. Classification and relation to age, occlusion, and concomitant injuries of teeth and teeth-supporting structures, and fractures of the mandibular body. Int J Oral Surg. 1977 Feb;6(1):12-21. doi: 10.1016/s0300-9785(77)80067-7. PMID 402318
- [Background] THOMA KH. Treatment of condylar fractures. J Oral Surg (Chic). 1954 Apr;12(2):112-20. No abstract available. PMID 13152606
- [Background] Zachariades N, Mezitis M, Mourouzis C, Papadakis D, Spanou A. Fractures of the mandibular condyle: a review of 466 cases. Literature review, reflections on treatment and proposals. J Craniomaxillofac Surg. 2006 Oct;34(7):421-32. doi: 10.1016/j.jcms.2006.07.854. Epub 2006 Oct 19. PMID 17055280
- [Background] Spiessl B, Schroll K. Gelenkfortsatz und gelenkkopfchenfracturen (Fractures of the condylar neck and head). Spezielle frakture und luxationslehre (Textbook of specialised fractures and dislocations) BD. I/I. Stuttgart: Thieme. 1972.
- [Background] Loukota RA, Neff A, Rasse M. Nomenclature/classification of fractures of the mandibular condylar head. Br J Oral Maxillofac Surg. 2010 Sep;48(6):477-8. doi: 10.1016/j.bjoms.2009.08.036. Epub 2009 Nov 6. No abstract available. PMID 19896755
- [Background] Chrcanovic BR. Open versus closed reduction: diacapitular fractures of the mandibular condyle. Oral Maxillofac Surg. 2012 Sep;16(3):257-65. doi: 10.1007/s10006-012-0337-6. Epub 2012 Jul 28. PMID 22842852
- [Background] He D, Yang C, Chen M, Bin J, Zhang X, Qiu Y. Modified preauricular approach and rigid internal fixation for intracapsular condyle fracture of the mandible. J Oral Maxillofac Surg. 2010 Jul;68(7):1578-84. doi: 10.1016/j.joms.2009.07.076. PMID 20430506
- [Background] Hlawitschka M, Eckelt U. Assessment of patients treated for intracapsular fractures of the mandibular condyle by closed techniques. J Oral Maxillofac Surg. 2002 Jul;60(7):784-91; discussion 792. doi: 10.1053/joms.2002.33246. PMID 12089693
- [Background] Molina CV, Moreno RO, Coloma OB, Meza VD, Silva MA. Preauricular approach: our alternative for surgical treatment of condylar fractures. International Journal of Oral and Maxillofacial Surgery. 2013;42:1236
- [Background] Mohan AP, Jeevan Kumar KA, Venkatesh V, Pavan Kumar B, Patil K. Comparison of preauricular approach versus retromandibular approach in management of condylar fractures. J Maxillofac Oral Surg. 2012 Dec;11(4):435-41. doi: 10.1007/s12663-012-0350-1. Epub 2012 Apr 4. PMID 24293937
- [Background] House JW. Facial nerve grading systems. Laryngoscope. 1983 Aug;93(8):1056-69. doi: 10.1288/00005537-198308000-00016. PMID 6877014
- [Background] House JW, Brackmann DE. Facial nerve grading system. Otolaryngol Head Neck Surg. 1985 Apr;93(2):146-7. doi: 10.1177/019459988509300202. No abstract available. PMID 3921901
- [Result] Rowe NL, Killey HC. Fractures of the facial skeleton: E. & S. Livingstone; 1955.
- [Result] Cascone P, Leonardi R, Marino S, Carnemolla ME. Intracapsular fractures of mandibular condyle: diagnosis, treatment, and anatomical and pathological evaluations. J Craniofac Surg. 2003 Mar;14(2):184-91. doi: 10.1097/00001665-200303000-00009. PMID 12621288
- [Result] Rowe NL, Killey HC. Fractures of the facial skeleton: Churchill Livingstone; 1968.
- [Result] Rowe NL. Surgery of the temporomandibular joint. Proc R Soc Med. 1972 Apr;65(4):383-8. doi: 10.1177/003591577206500438. No abstract available. PMID 5024527
- [Result] Al-Kayat A, Bramley P. A modified pre-auricular approach to the temporomandibular joint and malar arch. Br J Oral Surg. 1979 Nov;17(2):91-103. doi: 10.1016/s0007-117x(79)80036-0. PMID 298842
- [Result] Dolwick MF, Kretzschmar DP. Morbidity associated with the preauricular and perimeatal approaches to the temporomandibular joint. J Oral Maxillofac Surg. 1982 Nov;40(11):699-700. doi: 10.1016/0278-2391(82)90141-0. No abstract available. PMID 6957557
- [Result] Lima SM Jr, Asprino L, Moreira RW, de Moraes M. Surgical complications of mandibular condylar fractures. J Craniofac Surg. 2011 Jul;22(4):1512-5. doi: 10.1097/SCS.0b013e31821d4c6f. PMID 21778851
- [Result] Hall MB, Brown RW, Lebowitz MS. Facial nerve injury during surgery of the temporomandibular joint: a comparison of two dissection techniques. J Oral Maxillofac Surg. 1985 Jan;43(1):20-3. doi: 10.1016/s0278-2391(85)80008-2. PMID 3855313
- [Result] do Egito Vasconcelos BC, Bessa-Nogueira RV, da Silva LC. Prospective study of facial nerve function after surgical procedures for the treatment of temporomandibular pathology. J Oral Maxillofac Surg. 2007 May;65(5):972-8. doi: 10.1016/j.joms.2006.06.280. PMID 17448850
- [Result] Weinberg S, Kryshtalskyj B. Facial nerve function following temporomandibular joint surgery using the preauricular approach. J Oral Maxillofac Surg. 1992 Oct;50(10):1048-51. doi: 10.1016/0278-2391(92)90488-l. PMID 1527657
- [Result] Babakurban ST, Cakmak O, Kendir S, Elhan A, Quatela VC. Temporal branch of the facial nerve and its relationship to fascial layers. Arch Facial Plast Surg. 2010 Jan-Feb;12(1):16-23. doi: 10.1001/archfacial.2009.96. PMID 20083736
- [Result] Krayenbuhl N, Isolan GR, Hafez A, Yasargil MG. The relationship of the fronto-temporal branches of the facial nerve to the fascias of the temporal region: a literature review applied to practical anatomical dissection. Neurosurg Rev. 2007 Jan;30(1):8-15; discussion 15. doi: 10.1007/s10143-006-0053-5. Epub 2006 Nov 10. PMID 17096156
- [Result] Kim S, Matic DB. The anatomy of temporal hollowing: the superficial temporal fat pad. J Craniofac Surg. 2005 Sep;16(5):760-3. doi: 10.1097/01.scs.0000180010.83480.10. PMID 16192853
- [Result] Politi M, Toro C, Cian R, Costa F, Robiony M. The deep subfascial approach to the temporomandibular joint. J Oral Maxillofac Surg. 2004 Sep;62(9):1097-102. doi: 10.1016/j.joms.2003.10.013. PMID 15346360